CLINICAL TRIAL: NCT04638140
Title: Retrospective Assessment of the Morphology of Acetabular Defects: A 3D Reconstruction Approach
Status: Terminated | Type: Observational
Why Stopped: Inactive
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S61746
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hip Arthrosis; Hip Injuries
Keywords: Hip revision surgery
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy hip population
- Hip defect population

SUMMARY:
In this study, we aim to develop a statistical shape model and use it to reconstruct the shape of acetabula with severe defects (Paprosky 3a-3b). This will allow us to visualise and assess the morphology of the missing bone. In future studies we will use the obtained results to improve the design of acetabular implants for revision surgery.

ELIGIBILITY:
Trainings dataset for statistical shape model:

* Patients where a bilateral CT of the hip was performed with unilateral pathologies.
* We aim to include an equal amount of scans from each gender and varying ages.

Dataset of defect acetabula used for reconstruction:

* Patients who received a CT scan of the hip after removal of a primary/revision implant (e.g. patients where debridement was performed due to infection.)
* Patients where the defect can be classified as a Paprosky 3a or 3b defect.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Trainings dataset for statistical shape model:
  * Bones with irregularities, such as fractures or osteophytes
  * Patients who received radiation therapy in the past.
  * Patients with bone related diseases
  Dataset of defect acetabula used for reconstruction:
  • Patients who received radiation therapy in the past.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
3D morphology | 2 years
  Compare the 3D morphology of acetabular defects (missing bone) with traditional 2D classifications using CT images of patients with various degrees of bone defects.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leuven, Pellenberg, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No